CLINICAL TRIAL: NCT00291213
Title: Levetiracetam Treatment of Tardive Dyskinesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YaleHIC26585
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Levetiracetam

ARMS (2):
- Levetiracetram Administration (Experimental)
  Interventions: Drug: levetiracetam
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levetiracetam
  Arms: Levetiracetram Administration
Drug: placebo
  Arms: Placebo

SUMMARY:
This is a placebo-controlled study designed to learn if levetiracetam is effective for tardive dyskinesia.

ELIGIBILITY:
Inclusion Criteria: meet Glazer Morgenstern criteria for TD -

Exclusion Criteria: none

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Abnormal Involuntary Movement Scale (AIMS) Total Score | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Woods SW, Saksa JR, Baker CB, Cohen SJ, Tek C. Effects of levetiracetam on tardive dyskinesia: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2008 Apr;69(4):546-54. doi: 10.4088/jcp.v69n0405. PMID 18312060